CLINICAL TRIAL: NCT02613780
Title: iDesign Aberrometer for the Refractive Treatment of Early Keratoconus
Brief Title: Refractive Treatment of Early Keratoconus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150570-01H
Record Dates: First submitted 2015-11-17; First posted 2015-11-25 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Photorefractive Keratectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential group (Active Comparator): Photorefractive keratectomy will be performed 12-18 months after participants had crosslinking
  Interventions: Procedure: Crosslinking; Procedure: Photorefractive keratectomy; Device: iDesign® Advanced WaveScan Studio
- Simultaneous group (Active Comparator): Photorefractive keratectomy and crosslinking will be performed on the same day
  Interventions: Procedure: Crosslinking; Procedure: Photorefractive keratectomy; Device: iDesign® Advanced WaveScan Studio

INTERVENTIONS:
Procedure: Crosslinking — corneal collagen crosslinking with riboflavin
Procedure: Photorefractive keratectomy
Device: iDesign® Advanced WaveScan Studio — Used to map wavefront aberration in planning photorefractive keratectomy

SUMMARY:
Keratoconus is a bilateral, progressive corneal degenerative disorder that often leads to significant visual deterioration over time. Corneal collagen crosslinking with riboflavin (CXL) was developed as a treatment to halt the progression of keratoconus and thus negate the need for corneal transplantation. However, the treatment alone has little impact in terms of improving visual function. Photorefractive keratectomy (PRK) is the application of an excimer laser to treat a patient's refractive error, therefore decreasing the dependence on spectacles or contact lenses for improved vision.

Corneal collagen crosslinking combined with photorefractive keratectomy has been explored to partially correct the refractive error in keratoconic patients, whilst simultaneously stabilizing the corneal changes. Recently, the iDesign® Advanced WaveScan Studio (iDesign system; Abbot Medical Optics; Santa Ana, CA) has been launched as the most advanced high-resolution aberrometer. It is capable of mapping highly aberrated corneas for wavefront-guided laser procedures, and represents an important technological advance in treating corneal disease.

The purpose of this single center, prospective pilot study is to assess the safety and efficacy of combined wavefront-guided PRK and CXL in patients with early keratoconus using the iDesign® aberrometer. Results of this pilot study will be used to provide sample size estimates for an extension of the study, which aims to determine whether sequential or same day procedure leads to better outcomes.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the visual outcomes of combined wavefront-guided PRK and CXL in Krumeich stage 1 and 2 keratoconic eyes. The investigators will be conducting a prospective study at the University of Ottawa Eye Institute. A total of 24 patients will be enrolled in the study divided into two groups:

Group 1: PRK performed12-18 months after CXL; Group 2: PRK performed or on the same day as CXL

Participants will be followed at regular intervals for 1 year and information regarding visual, refractive, keratometric and higher order aberration outcomes will be collected.

The researchers aim to investigate the safety and efficacy of combined wavefront guided PRK and CXL. Results of this pilot study will used to provide estimates for sample size calculation for an extension of the study, which aims to determine whether sequential or same day procedure leads to better outcomes.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

1. Patients with confirmed diagnosis of keratoconus in Krumeich stage 1 or 2 who have received crosslinking 12-18 months prior, with follow up of at least 12 months

Group 2:

1. Diagnosis of keratoconus confirmed based on clinical examination findings and corneal topography
2. Evidence of progression of keratoconus occurring over the last 12 months defined as:

   i. An increase of maximum keratometry reading by 1 diopter or more (≥ 1 D), or ii. Evidence of clinical progression
3. Age between 21 and 60 years
4. Eyes satisfying all of Krumeich stage 1 or 2 criteria listed below i. Stage 1: eccentric corneal bulging, myopia, and/or astigmatism <5 D and corneal radius ≤48 D, no corneal opacities ii. Stage 2: myopia and/or astigmatism >5 D and <8 D and/or corneal radius ≤53 D, no central opacities, pachymetry ≥400 μm

Exclusion Criteria:

1. Age less than 21 years, or older than 60 years
2. Pregnant, or planning to become pregnant, or breastfeeding
3. Past history of Herpes Simplex Keratitis or corneal surgery (other than crosslinking)
4. Thin Cornea (<425 microns)
5. Other corneal disease, corneal scarring
6. History of chemical burns to the cornea or known healing problems
7. Known allergy to Riboflavin (vitamin B2)
8. If patient suffers from nystagmus or any other condition that would render it difficult for the patient to hold a steady gaze
9. Very advanced corneal ectasia (beyond Krumeich stage 2)
10. Poor visual potential
11. Vitamin C supplements within 1 week of the procedure
12. Lenticular changes (cataracts)
13. Programmed PRK treatment exceeding 50 microns in tissue depth

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in best-corrected visual acuity at followups | 1 year
  Best-corrected visual acuity (BCVA) will be measured in logMAR. Preoperative BCVA will be compared to BCVA postoperatively and at followups over 1 year using paired t tests.

SECONDARY OUTCOMES:
Intraoperative and postoperative complications | 1 year
  Number of patients with unexpected complications, as well as the type of complication will be collected over 1 year of followups.